CLINICAL TRIAL: NCT05314036
Title: Establishment of a Standard Operating Procedure for Screening of the Pathologies Associated With Prediabetes and Diabetes -The Wellness Transformation Network Pilot Study.
Brief Title: The Wellness Transformation Network Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SciMar Ltd. (Industry)
Collaborators: Source Nutraceutical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WTN-001
Record Dates: First submitted 2022-02-10; First posted 2022-04-06 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Non-Diabetic; Females Who Are Not Pregnant or Breast Feeding
Keywords: Glucose; Insulin; Prediabetes
MeSH Terms: conditions — Breast Feeding; Insulin Resistance; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acute Postprandial Blood Sampling (Experimental): Two-hour postprandial blood sampling following administration of a standardized test meal
  Interventions: Other: Standardized test meal

INTERVENTIONS:
Other: Standardized test meal — During this study visit, a standardized test meal will be administered. Blood samples will be collected at baseline and then every 30 minutes for 2 hours after test meal.

SUMMARY:
The purpose of the study is to establish a Standard Operating Procedure (SOP) for the screening of pathologies associated with prediabetes and type 2 diabetes.

DETAILED DESCRIPTION:
The proposed study will enable screening of pathologies associated with cardiometabolic diseases (i.e., hypertension, prediabetes, insulin resistance, diabetes, and obesity). The Meal-Induced Insulinemia and Glycemia (MIG) score will correlate with those dysfunctions that are components of the Absence of Meal-Induced Insulinemia (AMIS) syndrome. Overall the study aims:

1. To establish an SOP for screening pathologies associated with cardiometabolic diseases using a combination of biometrics and metabolomics.
2. To compare a participant's MIG score and hepatalin levels following consumption of a standardized test meal containing macronutrients, and the measurement of several indices of organ health associated with diabetes (i.e., body composition, handgrip strength, spirometry, blood pressure, and heart rate variability).

The study will involve 2 study visits: Visit 1 - Screening and Visit 2 - Intervention (Test meal administration and postprandial blood collection).

ELIGIBILITY:
Inclusion Criteria:

* Adults (males and females)18 years of age or older.
* Able to understand and communicate in English.
* Willing to answer a questionnaire on lifestyle and health status.
* Willing to undergo measurements of height, weight, waist circumference, hip circumference, blood pressure, heart rate and heart rate variability, body mass index, handgrip strength (handgrip dynamometry) testing, and pulmonary function (spirometry) testing.
* Willing to fast for 12 hours prior to two in-person study visits.
* Willing to consume a standardized test meal containing food ingredients.
* Willing to provide a urine sample.
* Willing to take a pregnancy test (female participants of childbearing potential).
* Willing to provide the research team with a listing of all current medications and Natural Health Products(NHPs).
* Willing to complete an online eDiary, including a 3-day food record.
* Willing to give blood samples (finger prick and blood sampling at defined intervals using an intravenous catheter)

Exclusion Criteria:

* Individuals diagnosed with diabetes.
* Women with confirmed pregnancy or who are breastfeeding.
* Individuals with allergy or sensitivity to any component of the standardized test meal (i.e., dextrose, lecithin, soy protein).
* Individuals with a fasting blood glucose of 7.0 mmol/L or higher.
* Individuals with abnormal glucose in their urine.
* Individuals who are related to or working for the clinic site, research staff, and study sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-01-17 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Establishment of proposed Wellness Transformation Network clinical trial procedures. | 2 Weeks
  Practical feasibility of the proposed Wellness Transformation Network clinical trial procedures (Yes/No)

SECONDARY OUTCOMES:
Time course and curve analysis of serum glucose response after the test meal administration. | Test: Baseline, every 30 minutes up to 2 hours after test meal administration
Time course and curve analysis of serum insulin response after the test meal administration. | Test: Baseline, every 30 minutes up to 2 hours after test meal administration
Time course and curve analysis of serum triglycerides response after the test meal administration. | Test: Baseline, every 30 minutes up to 2 hours after test meal administration
Time course and curve analysis of plasma hepatalin response after the test meal administration. | Test: Baseline, every 30 minutes up to 2 hours after test meal administration
Time course and curve analysis of Meal Induced Glycemia (MIG) scores response after the test meal administration. | Test: Baseline, every 30 minutes up to 2 hours after test meal administration
  MIG is calculated using the formula: MIG = (post meal insulin mIU/L X post meal glucose mmol/L) minus (fasted insulin mIU/L X fasted glucose mmol/L). Higher score equates to a worse (unhealthy) outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Vanu Ramprasath, PhD, Principal Investigator — Source Nutraceutical, Inc.
Locations (1):
- SNI Clinical Research, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No